CLINICAL TRIAL: NCT04596683
Title: Same-Day Discharge After Nipple-sparing Mastectomy or Skin-sparing Mastectomy With Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00000441
Record Dates: First submitted 2020-05-13; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Mastectomy; Lymphedema; Same Day Surgery; Nipple-sparing Mastectomy; Skin-sparing Mastectomy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — specific substance maruyama

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interested in SDS NSM or SSM (Experimental): Patients interested same day discharge after NSM or SSM that do not have conditions that would exclude them. Based on discharge outcome after surgery, will be split into SDS group and Admit group.
  Interventions: Procedure: Same-day NSM or SSM

INTERVENTIONS:
Procedure: Same-day NSM or SSM — Discharge home same-day after nipple-sparing mastectomy (NSM), or skin-sparing mastectomy (SSM)

SUMMARY:
This novel study will assess the feasibility and outcomes of same-day discharge following mastectomy with implant-based pre-pectoral reconstruction. This contrasts the current standard practice of admitting patients to the hospital as an inpatient for at least one night postoperatively. With the advent of pre-pectoral implant-based reconstructive techniques as opposed to the historical retro-pectoral breast reconstruction, patients experience significantly less post-operative pain, shorter recovery time, and improved mobility all of which support that patients lacking comorbidities are likely to meet discharge criteria the same day as surgery. Furthermore, advances in opioid sparing anesthesia and the Enhanced Recovery After Anesthesia protocol, has dramatically reduced pain scores and narcotic requirements after surgery at our institution. "Same day discharge" may reduce healthcare costs, decreases the risk of hospital-acquired infections and can increase patient satisfaction. Potential risks associated with same day discharge include readmissions, infections, limitations to pain management and other complications. The study will be conducted at MedStar System Hospitals and the population will be patients receiving pre-pectoral breast reconstruction following mastectomy that consent to the study. The project will be conducted as a prospective study where a carefully selected group of women without comorbidities undergoing mastectomy and pre-pectoral implant-based reconstruction will be offered same day discharge, educated about postoperative care preoperatively, be evaluated in the PACU and if they meet discharge criteria, will go home the same day as surgery. Those women who do not meet discharge criteria will stay overnight and be followed for outcomes, as well, as a comparison group. The primary endpoint for this study is patient satisfaction. Secondary outcomes include pain, complications including infection, hematomas, return to emergency room or urgent care, opiate equivalent use, and whether a patient would recommend same day discharge to others. Statistical analysis using means, 95% CI, frequency counts, descriptive statistics, fisher exact test and independent t-tests will evaluate differences between the same day discharge and admitted groups. Please see section 6 in the IRB protocol for more detail. We hypothesize that same day discharge provides acceptable patient satisfaction, pain control, complication rates with similar opiate equivalent use in comparison with overnight admission. Overall, we think this group will demonstrate positive outcomes on its own in these categories. We also believe that this study will demonstrate patients with same day discharge will recommend it to other women undergoing mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients either receiving nipple-sparing mastectomy or skin sparing mastectomy
* Patients with new diagnosis of cancer receiving mastectomy or those receiving mastectomy for preventative surgery
* Receiving implant-based pre-pectoral breast reconstruction
* Patients whose treatment is to be completed at MedStar System Hospitals
* Amenable to option of SDS prior to surgery
* Capable of giving informed consent

Exclusion Criteria:

* Active Smoker
* Patients with high risk comorbidities (significant cardiac disease, diabetes) that necessitate prolonged postoperative in house course

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-02-04 (Estimated); Study Completion 2022-02-04 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | Pre-op to Post-op Day 7
  Breast Q Survey Scores pre and post-op. All scores calculated on scale of 100 further divided into sections scored out of 100 analyzing psychosocial, physical, appearance, and care outcomes. Higher scores associated with better satisfaction.

SECONDARY OUTCOMES:
Complications | up to 30days post-op
  frequencies of infection, hematomas, return to emergency room or urgent care
Pain Scores | Preop to Post-op day 1
  American Pain Society Post-operative Outcome Survey pre and post-op surveys. Scored on basis of answers of 12 questions, divided into 5 categories of questions. Most composite category scores are associated with higher scores equaling poorer outcomes except for "perceptions of care" where higher scores demonstrate improved outcomes.

OTHER OUTCOMES:
Opioid use | Up to post-op day 20
  Post-op narcotic use recorded in log brought home by patients.Use to calculate average use per day after discharge and trends postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Eleni A Tousimis, MD, Principal Investigator — Medstar Georgetown Attending Physician
Locations (3):
- United States (3):
  - Medstar Georgetown University, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Medstar Franklin Square Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Alvarez IM, Tousimis EA. Reply: Breast Surgery in the Time of Global Pandemic: Benefits of Same-Day Surgery for Breast Cancer Patients Undergoing Mastectomy with Immediate Reconstruction during COVID-19. Plast Reconstr Surg. 2021 Aug 1;148(2):325e-326e. doi: 10.1097/PRS.0000000000008159. No abstract available. PMID 34228679